CLINICAL TRIAL: NCT03308929
Title: Prospective Multi-Center Clinical Evaluation Following Total Hip Arthroplasty With the G7 Dual Mobility System
Brief Title: Prospective G7 Dual Mobility Total Hip PMCF
Status: Active, not recruiting | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: H.CR.I.G.16.5
Record Dates: First submitted 2017-04-24; First posted 2017-10-13 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Clinical Outcomes; Functional Outcomes; Radiological Outcomes; Survivorship; Safety

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: G7 Dual Mobility hip — Total hip arthroplasty and implantation of the G7 device

SUMMARY:
This is a prospective multi-center clinical evaluation following recipients of the G7 Dual Mobility hip device. The primary objective is to characterize survivorship of the G7 hip at five years post-index procedure. Secondary objectives include documentation of clinical outcomes, safety and radiographic data.

DETAILED DESCRIPTION:
This multi-center prospective follow-up study will evaluate clinical outcomes, functional outcomes, radiological outcomes and further characterize the safety profile of the G7 Dual Mobility Hip Arthroplasty System. This will be accomplished by assessing these domains using the Harris Hip Score, UCLA Activity Score, and EQ-5D-3L, obtaining and assessing radiographs and the tracking of device or procedure related adverse events. Subjects will undergo unilateral primary or revision total hip arthroplasty and will then be followed for 10 years with intervals at 6 weeks, 1-, 2-, 3- 5- and 10 years. For the 10 year visit, subjects will not be required to present in their doctor's office, but will fill out a survey. Subsequent to 10 year data collection, the subject's participation in the study will be compete.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are undergoing revision hip arthroplasty

  -OR
* Patients who are undergoing total hip arthroplasty (THA) for the correction of a functional deformity

  - OR
* Patients in need of treatment of femoral neck fracture, and trochanteric fractures of the proximal femur with head involvement, unmanageable by other techniques

  - OR
* Patients suffer from substantial pain and/or limited function, are appropriate for a primary total hip arthroplasty, considered at high risk for dislocation and have one of the following:

  * Non-inflammatory degenerative joint disease, including osteoarthritis and avascular necrosis
  * Rheumatoid arthritis
* Decision to have a G7 Dual Mobility system implanted was made independently and prior to recruitment into study
* From 18 to 80 years of age (inclusive) at time of procedure
* BMI equal to or less than 35
* Unilateral total hip replacement
* Willing and able to comply with the study procedures

Exclusion Criteria:

* Patients undergoing total hip arthroplasty following non-union of previous surgically treated fracture.
* Infection, sepsis or osteomyelitis at the affected joint
* Significant osteoporosis as defined by treating surgeon
* Metabolic disorders which may impair bone formation
* Osteomalacia
* Distant foci of infections which may spread to the implant site
* Rapid joint destruction, marked bone loss or bone resorption on preoperative radiographs
* Underwent contralateral THA within 12 months of planned index procedure
* Contralateral THA planned within 12 months of index procedure
* Vascular insufficiency, muscular atrophy at the implant site or neuromuscular disease
* The patient is

  * A prisoner
  * A known alcohol or drug abuser
* The patient has any concomitant disease which is likely to jeopardize the functioning or success of the implant
* The patient is known to be pregnant
* The patient has a known sensitivity or allergy to one or more of the implanted materials, inducing but not limited to chromium, cobalt, and ceramic

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing revision hip arthroplasty, undergoing a hip arthroplasty to correct a functional deformity, patients seeking treatment for femoral neck fracture, and trochanteric fractures of the proximal femur with head involvement, unmanageable by other techniques, and patients with significant hip pain or functional limitations and who are at a high dislocation risk will be considered for the study. Patients may have avascular necrosis, osteo- or rheumatoid arthritis.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2017-02-28 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Survivorship of the study device | 5 years
  This is assessed by removal of the study device from the patient for any reason, including failure of the device, infection, or traumatic injury.

SECONDARY OUTCOMES:
Radiographic measurements of the implanted device | 10 years
  Standard AP radiographs of implanted hip will assess the positioning of the device as well as lucencies and other potential anomalies.
Frequency and incidence of adverse events for all subjects with particular focus on those related or potentially related to the device | 10 years
  Assessed by tracking the type of adverse event, severity and relation of the event(s) to the study device
Patient Physical Activity | 10 years
  UCLA activity score - patient self assessment
Patient Quality of Life | 10 years
  EQ-3L-5D quality of life measure - patient self assessment
Harris Hip Score | 10 years
  Harris Hip score measures pain, function, absence of deformity, and range of motion. Scores range from 0-100 with higher scores representing less dysfunction and better outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Hillary Overholser, MS, Study Director — Zimmer Biomet
Locations (6):
- United States (6):
  - Jersey City Medical Center, Jersey City, New Jersey
  - New Mexico Orthopaedics, Albuquerque, New Mexico
  - University of North Carolina, Chapel Hill, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Tidewater Orthopaedics, Hampton, Virginia
  - Ortho Virginia, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Undecided